CLINICAL TRIAL: NCT05182177
Title: A Multi-Center, Retrospective Review of Implant-Based Post Mastectomy Breast Reconstruction Utilizing SurgiMend® Collagen Matrix in Prepectoral and Submuscular Surgical Approaches
Brief Title: The SurgiMend PRS Retrospective Study
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: T-SUPORT-001
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Reconstructive Surgical Procedures
Keywords: breast reconstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SurgiMend PRS — SurgiMend® PRS and SurgiMend® PRS Meshed are intended for implantation to reinforce soft tissue where weakness exists and for surgical repair of damaged or ruptured soft tissue membranes. SurgiMend® PRS and SurgiMend® PRS Meshed are specifically indicated for plastic and reconstructive surgery, including breast reconstruction.
  Other Names: SurgiMend PRS Meshed

SUMMARY:
The SurgiMend® PRS Retrospective Study will evaluate the performance and safety of SurgiMend® PRS and SurgiMend® PRS Meshed when used for soft tissue reinforcement under the product's indications for use.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has reviewed the ethics-approved consent form and has provided consent for data collection
2. Subject is a female over the age of 18 at the time of index surgery (mastectomy)
3. Subject had mastectomy performed for cancer or as a cancer prophylaxis
4. The surgical plan included one of the following approaches:

   1. Immediate unilateral or bilateral prepectoral DTI or TE/I breast reconstruction following nipple-sparing, skin-sparing, or skinreducing mastectomy with the use of SurgiMend® PRS or SurgiMend® PRS Meshed
   2. Immediate unilateral or bilateral submuscular DTI or TE/I breast reconstruction following nipple-sparing, skin-sparing, or skin-reducing mastectomy with the use of SurgiMend® PRS or SurgiMend® PRS Meshed
5. If subject received bilateral breast reconstruction, the subject must have received the same surgical technique for both breasts including the implantation of SurgiMend® PRS or SurgiMend® PRS Meshed
6. If subject received unilateral breast reconstruction, there was no surgical intervention on the contralateral breast within 12 months post-operatively
7. Subject underwent mastectomy (index surgery) at a minimum of 24 months prior to study initiation at site

Exclusion Criteria:

1. The surgical plan included muscle flaps to supplement the breast mound
2. The reconstruction plan included hybrid implant coverage with another type of mesh (e.g., use of another mesh or ADM in addition to SurgiMend®)
3. Subject had received prior breast augmentation, mastopexy, or breast reduction surgeries (does not include breast biopsy)
4. Subject was a user of any nicotine products (cigarettes, chewing tobacco, vapor, etc.) (within 6 weeks before index surgery)
5. Subject had uncontrolled Type I or Type II diabetes (HbA1C >9)
6. Subject had previously undergone radiation therapy to the chest wall prior to index surgery
7. Subject had been diagnosed with advanced stage disease (stage 3 or 4, or inflammatory cancer)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data will be collected for 50 female subjects that have been implanted with SurgiMend® PRS and 50 female subjects that have been implanted with SurgiMend® PRS Meshed according to the IFU.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Performance of SurgiMend | 24 months
  The primary endpoint of this study is the proportion of patients who did not require additional surgical interventions at or associated with the site of the original reconstruction within 12 months after SurgiMend® PRS or SurgiMend® PRS Meshed implantation.

SECONDARY OUTCOMES:
Safety of SurgiMend | 24 months
  The secondary endpoint of this study is the occurrence of relevant (S)AEs within 12 months of SurgiMend® PRS or SurgiMend® PRS Meshed implantation.

CONTACTS AND LOCATIONS:
Locations (6):
- AULSS9 Scaligera, Verona, Veneto, Italy
- Ospedale Regionale di Lugano; Sede Ospedale Italiano, Viganello, Switzerland
- United Kingdom (4):
  - Royal Free Hospital, London, North West
  - Royal Hallamshire Hospital, Sheffield, Yorkshire
  - Guy's and St Thomas' NHS Foundation Trust, London
  - North Manchester General Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Undecided